CLINICAL TRIAL: NCT03031561
Title: Breast Microcalcifications Identified With MicroPure as a Marker for Malignancy Compared to Grayscale Ultrasound and Mammography (Using Biopsy as the Reference Standard)
Brief Title: Ultrasound Imaging Technique in Detecting Breast Microcalcifications in Patients Undergoing Biopsy for a Breast Abnormality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 12D.17; JT 1962 (Other: JeffTrial Number)
Record Dates: First submitted 2017-01-20; First posted 2017-01-25 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma; Microcalcification
MeSH Terms: conditions — Breast Neoplasms; Calcinosis | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (standard ultrasound, MicroPure, biopsy) (Experimental): Patients undergo grayscale and MicroPure ultrasound imaging followed by sonographic or stereotactic guided core needle biopsy or surgical resection. Surgical specimens are then x-rayed.
  Interventions: Device: Ultrasound; Device: MicoPure ultrasound; Procedure: Biopsy of Breast

INTERVENTIONS:
Device: Ultrasound — Undergo standard ultrasound
  Other Names: Ultrasound Imaging; US
Device: MicoPure ultrasound — Undergo MicoPure ultrasound
Procedure: Biopsy of Breast — Undergo breast biopsy or surgical resection
  Other Names: Breast Biopsy

SUMMARY:
This clinical trial studies a new type of ultrasound technique, MicroPure, in detecting breast microcalcifications in patients undergoing biopsy for a breast abnormality. Ultrasound sends sound waves into the body, and the sound waves reflected back are interpreted by the machine into a grayscale image. MicroPure uses a filter that adjusts the brightness and gives color to the ultrasound images, which may allow doctors to better identify microcalcifications. Microcalcifications are tiny deposits of calcium in the breast that cannot be felt but can be detected by imaging. A group of microcalcifications may indicate that cancer is present.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate MicroPure relative to grayscale ultrasound imaging for the identification of microcalcifications with mammography as the reference standard.

SECONDARY OBJECTIVES:

I. Evaluate MicroPure compared to grayscale ultrasound imaging and mammography for the characterization of breast abnormalities associated with microcalcifications using biopsy results as the reference standard (sensitivity and specificity will be calculated).

II. Evaluate MicroPure relative to specimen x-ray imaging for the identification of breast microcalcifications with pathology as the reference standard.

III. Estimate the improvements in patient care that may be achievable if MicroPure guided core needle biopsy procedures can replace some surgical excisions for the evaluation of breast abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent
* Be scheduled for a sonographic or stereotactic guided core needle biopsy or surgical excision for the evaluation of a breast lesion or abnormality containing microcalcifications seen on mammography

Exclusion Criteria:

* Is clinically unstable, severely ill, or moribund

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Number of microcalcifications seen on MicroPure ultrasound | Baseline
  The number of microcalcifications seen on MicroPure ultrasound will be recorded and compared to x-ray imaging of the area undergoing the biopsy procedure (as the reference standard). The difference in agreement between the two ultrasound modes (relative to mammography) will be assessed using McNemar's test for correlated proportions, where p-values less than 0.05 are considered significant. A dichotomous parameters indicating agreement with mammography with respect to the exact number of microcalcifications (as yes or no) will be calculated and compared.
Number of microcalcifications seen on grayscale ultrasound | Baseline
  The number of microcalcifications seen on grayscale ultrasound will be recorded and compared to x-ray imaging of the area undergoing the biopsy procedure (as the reference standard). The difference in agreement between the two ultrasound modes (relative to mammography) will be assessed using McNemar's test for correlated proportions, where p-values less than 0.05 are considered significant. A dichotomous parameters indicating agreement with mammography with respect to the exact number of microcalcifications (as yes or no) will be calculated and compared.

SECONDARY OUTCOMES:
Number of microcalcifications determined by pathology findings | Baseline
  The results of the three imaging methods will be compared to the pathology findings using the American College of Radiology Breast Imaging Reporting and Data System lexicon for the assessment of breast lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Forsberg, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/